CLINICAL TRIAL: NCT03046004
Title: The Effect of Receiving Information About the Benefits and Harms of Mammography Screening on Women's Decision Making
Brief Title: Effect of Information About the Benefits and Harms of Mammography on Women's Decision Making
Acronym: InforMa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Hospital del Mar (Other); Canary Islands Health Service (Unknown); Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Montserrat Rue, Professor, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI14/00113
Record Dates: First submitted 2017-02-04; First posted 2017-02-08 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer Screening
Keywords: breast cancer; screening; decision aid; informed choice; decisional conflict
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid (Experimental): Women in the intervention arm will receive a leaflet with detailed information on the benefits (breast cancer mortality reduction, less intensive treatments) and harms (false positive results and overdiagnosis).
  Interventions: Other: Decision aid for breast cancer screening
- Control (Active Comparator): Women in the control arm will receive a standard leaflet that does not mention harms and recommends accepting the invitation to participate in the biennial exams of the EDBCP.
  Interventions: Other: Standard leaflet

INTERVENTIONS:
Other: Decision aid for breast cancer screening — Women in the intervention arm will receive a leaflet with detailed information on the benefits (breast cancer mortality reduction, less intensive treatments) and harms (false positive results and overdiagnosis).
  Arms: Decision aid
Other: Standard leaflet — Women in the control arm will receive a standard leaflet that does not mention harms and recommends accepting the invitation to participate in the biennial exams of the EDBCP.
  Arms: Control

SUMMARY:
The aim of this study is to assess the effect of receiving information about the benefits and harms of mammography screening on informed choice, decisional conflict, intention to participate in the Early Detection of Breast Cancer Program (EDBCP), and satisfaction. The primary outcome is informed choice about breast screening (adequate knowledge, and consistency between attitudes and intentions). The sample of participants is composed by 400 women from Catalonia and the Canary Islands (Spain) who will receive their first invitation to participate in the EDBCP of the Public Health Service in a period of 2-4 months.

DETAILED DESCRIPTION:
The selected women will receive a letter of invitation with information about the study. In the following 1-2 weeks they will receive a phone call to confirm that they have received the mailed letter and to assess the inclusion criteria. If they agree to participate in the study, they will be asked for informed consent. All the participants will receive a first questionnaire, the pre-intervention survey (10-15 minutes), via web or regular mail. Trained interviewers will collect the responses by phone for women who prefer this method. Once the pre-intervention survey is completed, women will receive the leaflet (intervention or control) via regular mail. Two weeks later, the participants will be contacted again to collect the post-intervention survey (15-20 minutes), via web or by phone. Participation in the mammographic exams of the EDBCP will be collected in the three-month period following the corresponding invitation letter.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 49-50 who - in 2-4 months - will be invited to participate for the first time in the EDBCP of the Institut Hospital del Mar d'Investigacions Mèdiques (IMIM, Barcelona), ICO-Hospitalet (Hospitalet de Llobregat), Lleida Health Region, and the Canary Islands.
* Women with low health literacy will be included

Exclusion Criteria:

* Previous history of breast cancer
* Difficulty speaking Spanish or Catalan
* Cognitive impairment to understand or complete the materials based on the interviewer judgment

Ages: 49 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Informed choice | Two weeks after the intervention
  The primary outcome is informed choice about breast screening (adequate knowledge, and consistency between attitudes and intentions). See Hersch 2015.

SECONDARY OUTCOMES:
Breast screening attitudes | Two weeks after the intervention
  According to Hersch 2015
Breast screening intention | Two weeks after the intervention and after being invited to be screened
  According to Hersch 2015
Decisional conflict | Two weeks after the intervention
  According to Hersch 2015
Confidence in the decision made | Two weeks after the intervention
  According to Hersch 2015
Anxiety about screening participation | Two weeks after the intervention
  According to Hersch 2015
Worry about breast cancer | Two weeks after the intervention
  According to Hersch 2015
Anticipated regret | Two weeks after the intervention
  According to Hersch 2015
Time perspective | Two weeks after the intervention
  According to Hersch 2015
Perceived importance of benefit/harms of screening | Two weeks after the intervention
  According to Hersch 2015
Perceived risk of breast cancer | Two weeks after the intervention
  According to Hersch 2015

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Rué, PhD, Principal Investigator — Universitat de Lleida-IRBLLEIDA
Locations (1):
- Lleida Biomedical Research Institute (IRBLLEIDA), Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toledo-Chavarri A, Rue M, Codern-Bove N, Carles-Lavila M, Perestelo-Perez L, Perez-Lacasta MJ, Feijoo-Cid M; InforMa Study Group. A qualitative study on a decision aid for breast cancer screening: Views from women and health professionals. Eur J Cancer Care (Engl). 2017 May;26(3). doi: 10.1111/ecc.12660. Epub 2017 Feb 1. PMID 28145105
- [Background] Perez-Lacasta MJ, Martinez-Alonso M, Garcia M, Sala M, Perestelo-Perez L, Vidal C, Codern-Bove N, Feijoo-Cid M, Toledo-Chavarri A, Cardona A, Pons A, Carles-Lavila M, Rue M; with the InforMa Group. Effect of information about the benefits and harms of mammography on women's decision making: The InforMa randomised controlled trial. PLoS One. 2019 Mar 26;14(3):e0214057. doi: 10.1371/journal.pone.0214057. eCollection 2019. PMID 30913217
- [Background] Pons-Rodriguez A, Martinez-Alonso M, Perestelo-Perez L, Garcia M, Sala M, Rue M; en nombre del grupo InforMa; El grupo InforMa esta formado por. [Informed choice in breast cancer screening: the role of education]. Gac Sanit. 2021 May-Jun;35(3):243-249. doi: 10.1016/j.gaceta.2020.01.002. Epub 2020 Mar 12. Spanish. PMID 32173050
- [Result] Hersch J, Barratt A, Jansen J, Irwig L, McGeechan K, Jacklyn G, Thornton H, Dhillon H, Houssami N, McCaffery K. Use of a decision aid including information on overdetection to support informed choice about breast cancer screening: a randomised controlled trial. Lancet. 2015 Apr 25;385(9978):1642-52. doi: 10.1016/S0140-6736(15)60123-4. Epub 2015 Feb 18. PMID 25701273
- [Derived] Carles M, Martinez-Alonso M, Pons A, Perez-Lacasta MJ, Perestelo-Perez L, Sala M, Vidal C, Garcia M, Toledo-Chavarri A, Codern N, Feijoo-Cid M, Romero A, Pla R, Soler-Gonzalez J, Castells X, Rue M; InforMa Group. The effect of information about the benefits and harms of mammography on women's decision-making: study protocol for a randomized controlled trial. Trials. 2017 Sep 12;18(1):426. doi: 10.1186/s13063-017-2161-7. PMID 28899412